CLINICAL TRIAL: NCT07160153
Title: Cannabis Abstinence and Neurocognitive Assessment in Adolescence
Acronym: CANAA
Status: Recruiting | Type: Observational
Sponsor: University Hospital Pilsen (Other)
Responsible Party: Sponsor
Other Study IDs: CANAA
Record Dates: First submitted 2025-08-27; First posted 2025-09-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Cannabis Dependence; Harmful Use; Cognitive Assessment
Keywords: Cannabis Dependence; Cannabis Use Disorder; Abstinence; Cognitive Function; Disorder; Abstinence; Cognitive Function; Neuropsychological
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Adolescents aged 15-18 years with a diagnosis of cannabis dependence or harmful cannabis use.
  Interventions: Diagnostic Test: Neurocognitive assessment; Diagnostic Test: Urine toxicological assessment

INTERVENTIONS:
Diagnostic Test: Neurocognitive assessment — Neurocognitive battery:
  TMT-Trail Making Test Auditory Verbal Learning Test Stroop Test Tower of London (ToL), Shallice version Continuous Performance Test-Identical Pairs
  Other psychometrics:
  The level of dependence is quantified using the CAST (Cannabis Abuse Screening Test)
Diagnostic Test: Urine toxicological assessment — Urine toxicological assessment

SUMMARY:
Cannabis Abstinence and Neurocognitive Assessment in Adolescence

DETAILED DESCRIPTION:
Evaluate the development of cognitive functions following attainment of abstinence in a group of adolescents with cannabis dependence or harmful cannabis use. Abstinence is confirmed by toxicological testing.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 15-18 years with a diagnosis of cannabis dependence or harmful cannabis use.

Exclusion Criteria:

* psychiatric comorbidity - Dual diagnosis, including psychotic disorders, mood disorders, severe organic brain damage, or autism spectrum disorder, with the exception of compensated and stabilized anxiety disorder. Psychopharmacological treatment is permitted, except for antipsychotics prescribed for psychosis.
* somatic comorbidity - Severe endocrine disorders such as diabetes mellitus, thyroid dysfunction, or severe cardiovascular disease.
* Violation of abstinence between the first and second neuropsychological assessments, as well as severe decompensation of mental state requiring modification of established psychopharmacological treatment.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents aged 15-18 years with a diagnosis of cannabis dependence or harmful cannabis use.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in performance TMT-B | 8 weeks
  Change in performance on the Trail Making Test - Part B (TMT-B) [Time Frame: after 8 weeks of abstinence from cannabis]

SECONDARY OUTCOMES:
Change in performance on AVLT | 8 weeks
  Change in performance on the Auditory Verbal Learning Test (AVLT) [Time Frame: after 8 weeks of abstinence]
Change in performance on the Stroop Test | 8 weeks
  Change in performance on the Stroop Test [Time Frame: after 8 weeks of abstinence]
Change in performance on the Tower of London | 8 weeks
  Change in performance on the Tower of London (Shallice version) [Time Frame: after 8 weeks of abstinence]
Change in performance on CPT-IP | 8 weeks
  Change in performance on the Continuous Performance Test - Identical Pairs (CPT-IP) [Time Frame: after 8 weeks of abstinence]

OTHER OUTCOMES:
Cannabis Abuse Screening Test versus degree of neurocognitive impairment | 8 weeks
  Correlation between severity of cannabis dependence (Cannabis Abuse Screening Test, CAST) and degree of neurocognitive impairment [Time Frame: baseline and after 8 weeks of abstinence]

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Pilsen, Pilsen, Czechia, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet because we are still recruiting and waiting for primary outcome.